CLINICAL TRIAL: NCT07338669
Title: Hamburg Acute Renal Injury Study
Brief Title: Hamburg Acute Renal Injury Study (HARIS)
Acronym: HARIS
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV6037-4337-BO-ff HARIS
Record Dates: First submitted 2025-12-07; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury; Acute Kidney Injury (AKI)
Keywords: Acute Kidney Injury; AKI; Prospective observational cohort study
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — plasma (EDTA), serum, blood cells, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI group: Group consists of adult hospitalized individuals, who meet the 2012 Kidney Disease: Improving Global Outcomes (KDIGO) criteria for acute kidney injury (AKI). Participants will be prospectively followed for clinical course, kidney function, biomarker analysis, and outcomes. No experimental interventions are performed. All care follows standard clinical practice.
- Control group: Group consists of adult hospitalized individuals with an acute illness, who have not developed acute kidney injury (AKI). Participants will be prospectively followed for clinical course, kidney function, biomarker analysis, and outcomes. No experimental interventions are performed. All care follows standard clinical practice.

SUMMARY:
The Hamburg Acute Renal Injury Study (HARIS) is a prospective observational cohort study aimed at investigating the mechanisms, risk factors, and clinical determinants of acute kidney injury (AKI) trajectories and consequences.

DETAILED DESCRIPTION:
The Hamburg Acute Renal Injury Study (HARIS) is a prospective observational cohort study that includes hospitalized adults (≥18 years) at the time of acute kidney injury (AKI). Potential participants are identified during hospital care, and a structured IT-supported clinical screening system helps detect AKI cases in real time. In parallel, a control group of hospitalized adults with acute illness who have not developed AKI is enrolled to enable comparative analyses of specific risk factors, pathophysiology, and outcomes. All participants undergo a standardized clinical assessment of kidney function, comorbidities, hemodynamic status, medication exposure, procedures, and laboratory parameters. The study includes serial collection of clinical data and biosamples (blood and urine) at study inclusion, during hospitalization, and at 3-month after discharge. All biospecimens are processed within a harmonized pipeline and stored in the Hamburg and European Renal Omics-Biobank (HERO). Beyond the identification of clinical determinants of AKI trajectories, the central objective of HARIS is to identify biological pathways of sustained kidney injury and repair, improve risk stratification, evaluated prognostic biomarkers, and support the development of precision medicine approaches in post AKI care. Long-term outcomes including progressive chronic kidney disease, cardiovascular events, hospital readmissions, and mortality are collected through annual structured follow-ups. No experimental interventions are performed and all clinical management follows standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized individuals with acute kidney injury (AKI), defined by the 2012 Kidney Disease: Improving Global Outcomes (KDIGO) criteria or hospitalized individuals with acute illness who have not developed AKI (control group)
* Age ≥ 18 years at time of enrollment
* Personally signed informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized individuals with acute kidney injury (AKI) or at risk for AKI will be identified during routine medical care and invited for study participation. Routine clinical identification of AKI includes an IT-based screening system.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Kidney Function Recovery after AKI | assessed at discharge, 3-months after discharge, and annual follow-up
  Improvement of kidney function after acute kidney injury, defined by partial or complete return of the kidney function toward baseline values
Persistent Kidney Function Decline | assessed at discharge, 3-months after discharge, and annual follow-up
  Sustained impairment of kidney function following acute kidney injury, characterized by incomplete recovery and persistently reduced kidney function over follow-up.
Development or Progression of Chronic Kidney Disease | assessed at 3-months after discharge, and annual follow-up
  New onset or worsening of chronic kidney disease during follow-up, assessed based on changes in kidney function over time.
End-stage kidney disease (ESKD) | assessed at discharge, 3-months after discharge, and annual follow-up
  Occurrence of ESKD, characterized by the initiation of maintenance kidney replacement therapy, kidney transplantation or a persistent eGFR < 15 ml/min/1.73m2
Renal mortality | assessed at discharge, 3-months after discharge, and annual follow-up
  Death attributable to kidney-related causes as determined by medical record review.
Cardiovascular Outcomes | assessed at discharge, 3-months after discharge, and annual follow-up
  cardiovascular death, myocardial infarction, heart failure, arrhythmia, stroke

SECONDARY OUTCOMES:
Incidence of vascular diseases | assessed at discharge, 3 months after discharge, and annual follow-up
  Occurrence of vascular disease, including coronary artery disease, peripheral artery disease, or cerebrovascular disease after AKI
Incidence of Dementia | assessed at discharge, 3 months after discharge, and annual follow-up
  New diagnosis of dementia occurring during follow-up after AKI
Incidence of Cancer | assessed at discharge, 3 months after discharge, and annual follow-up
  New diagnosis of malignant disease occurring during follow-up after AKI
Incidence of Infections | assessed at discharge, 3 months after discharge, and annual follow-up
  New diagnosis of infections occurring during follow-up after AKI
Incidence of psychosomatic or Psychiatric Disorders | assessed at discharge, 3 months after discharge, and annual follow-up
  New diagnosis of psychosomatic or psychiatric disorders occurring during follow-up after AKI

CONTACTS AND LOCATIONS:
Overall Officials: Tobias B Huber, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany